CLINICAL TRIAL: NCT03344809
Title: ENABLE-NGS: Enhancing Diagnosis in Chronic B-cell Lymphoproliferative Disorders Using Next-Generation Sequencing
Brief Title: Enhancing Diagnosis in Chronic B-cell Lymphoproliferative Disorders Using Next-Generation Sequencing
Acronym: ENABLE-NGS
Status: Active, not recruiting | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR4383
Record Dates: First submitted 2017-02-07; First posted 2017-11-17 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Lymphoma
Keywords: lymphoma; unclassifiable; next; generation; sequencing
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * 20mls of PB in EDTA
  * Further 20mls PB in EDTA in cases where the first sample does not yield adequate DNA.
  * 5ml of BM in EDTA (optional for patients not undergoing bone marrow as part of normal work-up.
Oversight: Data Monitoring Committee: No

SUMMARY:
To enhance the diagnosis of unclassifiable, non-CLL B-LPDs using next-generation sequencing technology.

DETAILED DESCRIPTION:
In recent years, next generation sequencing has revealed the genomic landscape of lymphoid disorders and identified mutations that have improved our understanding of their pathogenesis. It has also revealed new targets for drug development. While some of these mutations, such as the BRAF V600E mutation in Hairy Cell Leukaemia (HCL)2, are now accepted as disease defining mutations, others such as MYD88 and NOTCH1/2 mutations are found in more than one subtype of B-LPD3. The overlapping nature of some of these molecular aberrations could have important implications for treatment of these disorders as we move towards targeted therapy. EZH2 inhibitors, which are currently in early phase trials, are one such example of targeted therapy for B-LPDs based on mutations identified by next generation sequencing (NGS)4. The genetic makeup of these tumours is also likely to influence future classification systems.

At present, an integrated approach incorporating morphology and immunophenotyping remains integral to the classification of B-LPDs. The Haemato-oncology department at the Royal Marsden Hospital has an international reputation in the development of immunophenotyping as a tool for the diagnosis of lymphoproliferative disorders. For example, the CLL score developed by the Haemato-Oncology department continues to be used in several centres around the world for the diagnosis of CLL5. A similar score proposed for HCL by our Haemato-Oncology department is also widely used (6). On a service evaluation, we found 100% concordance between a HCL score of 4 and presence of the BRAF mutation in samples referred to us (unpublished data).

Our plan therefore is to systematically study unclassifiable groups of B-LPD by creating a well-defined immunomorphology work flow for their identification. Samples thus identified will be screened using a next-generation sequencing (NGS) panel which is able to detect well established, B-LPD associated translocations and genetic mutations.

ELIGIBILITY:
Inclusion Criteria:

* Chronic, mature clonal B-cell malignancy that is not assignable to a specific WHO category by current technology (see flowchart in section below).

Exclusion Criteria:

* Non-clonal B-cell proliferation.
* High grade and/or immature clonal B-cell malignancy.
* Bone marrow samples with less than 20% infiltration will be excluded
* Samples from patients with a known classifiable chronic B-LPD based on lymph node biopsy for e.g. staging bone marrow samples on a patient with marginal zone lymphoma. If a definitive diagnosis is established on a subsequent lymph node biopsy, patient will remain on study and this will be correlated with NGS findings.
* Patient unable to provide consent for tumour and germ line samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering with an unclassifiable B-cell lymphoproliferative disorder
Sampling Method: Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2016-08; Primary Completion 2023-04 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of cases where a definite category and/or detectable mutation can be identified. | 2 years
  This will be reported as a percentage of the total number of cases sequenced

SECONDARY OUTCOMES:
Demographics and distribution in each immunomorphological category | 2 years
  Age and sex distribution will be reported along with the proportion of cases in each immunomorphologic category
Correlation of each immunomorphological category with the mutation profile. | 2 years
  The distribution of mutations within each immunomorphological category will be reported descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Iyengar, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom